CLINICAL TRIAL: NCT01955135
Title: DECREASING THE NEED FOR MECHANICAL VENTILATION AFTER RETINOPATHY OF PREMATURITY SURGERY: Sedation vs General Anesthesia
Brief Title: Anesthesia for Retinopathy of Prematurity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, assistant professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010 /145
Record Dates: First submitted 2013-09-04; First posted 2013-10-07 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Retinopathy
Keywords: Prematurity, Retinopathy, propofol, ketamine, sedation
MeSH Terms: conditions — Retinal Diseases; Premature Birth | interventions — Ketamine; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sedation (Active Comparator): The sedation group (Group S, n=30), received 1 mg/kg ketamine and 1 mg/kg propofol as a bolus for induction. The patients then received an infusion of 100-150 mcg/kg/min propofol and 0.25mg/kg/h of ketamine for maintenance.
  Interventions: Drug: Ketamine; Drug: propofol
- general anesthesia (Active Comparator): In the general anesthesia group (Group G, n=30), anesthesia was induced using 8% sevoflurane by inhalation with 50% nitrous oxide in oxygen; endotracheal intubation was facilitated without use of a neuromuscular blocker agent. Anesthesia was maintained with sevoflurane (2%) and 50% nitrous oxide in oxygen.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Ketamine — 1mg/kg bolus intravenous, 0.25mg/kg/hour intravenous for maintenance of sedation
  Other Names: ketalar, 50mg/ml
  Arms: sedation
Drug: Sevoflurane — anesthesia was induced using 8% sevoflurane by inhalation with 50% nitrous oxide in oxygen; Anesthesia was maintained with sevoflurane (2%) and 50% nitrous oxide in oxygen
  Other Names: sevorein
  Arms: general anesthesia
Drug: propofol — 1 mg/kg propofol as a bolus for induction. The patients then received an infusion of 100-150 mcg/kg/min propofol
  Other Names: pofol
  Arms: sedation

SUMMARY:
Premature infants experience more respiratory problems after surgical procedures. The investigators aimed to compare general anesthesia with sedation on the need for post-operative mechanical ventilation in infants undergoing retinopathy of prematurity surgery.

DETAILED DESCRIPTION:
60 patients who underwent laser surgery due to retinopathy of prematurity (ROP) were included in the study. The sedation group (Group S, n=30), received 1 mg/kg ketamine and 1 mg/kg propofol as a bolus for induction. The patients then received an infusion of 100-150 mcg/kg/min propofol and 0.25mg/kg/h of ketamine for maintenance. In the general anesthesia group (Group G, n=30), anesthesia was induced using 8% sevoflurane by inhalation with 50% nitrous oxide in oxygen; endotracheal intubation was facilitated without use of a neuromuscular blocker agent. Anesthesia was maintained with sevoflurane (2%) and 50% nitrous oxide in oxygen. Our primary objective was to evaluate the need for post-operative mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* infants aged 32-40 weeks who were scheduled to undergo laser surgery for treatment of ROP

Exclusion Criteria:

* The exclusion criteria were patients requiring inotropic support,
* the need for mechanical ventilation or intubation in the 3 days prior to the operation,
* known allergy or hypersensitivity reaction to ketamine and propofol,
* age ˃40 weeks.

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Respiratory failure after retinopathy of prematurity surgery in premature infants. | 1 Day (From end of anaesthesia till discharge from the recovery room )
  Most of premature infants have chronic lung disease, for this reason endotracheal intubation causes some problems, because they have irritable airway. Administration of sedation and avoiding endotracheal intubation can be better for postsurgical outcomes.
  How many infants needed endotracheal intubation and mechanical ventilation were recorded.

SECONDARY OUTCOMES:
Blood Pressure | 1 Day (From start of anaesthesia till discharge from the operation room)
  non invasive blood pressure measured
Heart rate | 1 Day (From start of anaesthesia till discharge from the recovery room )
  heart rate per minute were recorded

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE ÜLGEY, MD, Study Director — TC Erciyes University